CLINICAL TRIAL: NCT05101174
Title: Effects of an Integrated Intervention Program on Neurocognition in Late-Middle-Aged and Older Adults Relative to ApoE Genotypes: An ERP Study
Brief Title: Exercise and Neurocognition in Adults Relative to ApoE Genotype
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Yu-Kai Chang, Professor, National Taiwan Normal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PACNL_IIP and Neurocog_ERP
Record Dates: First submitted 2021-09-26; First posted 2021-11-01 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Exercise Training; Neurocognitive Function; Aging
Keywords: physical fitness; meditation; social interaction; Apolipoprotein E; aging; event-related potential
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Intervention Group (IIG) (Experimental): The IIG attends 150 min exercise per week, which consists of one 90-min trainer-supervised program and multiple online sessions, for 6 months.
  Intervention: aerobic exercise, resistance exercise, coordinative exercise, flexibility, social interaction, and meditation.
  Interventions: Behavioral: Integrated Intervention Group (IIG)
- Control Group (Other): The control group is invited to attend one 60-min online educational course per week for 6 months.
  Intervention: 60-min online educational program.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Integrated Intervention Group (IIG) — The IIG attends 150 min exercise per week, which consists of one 90-min trainer-supervised session and multiple online sessions for 6 months. Each session consists of (1) warm-up, (2) resistance exercise and flexibility exercise, (3) resistance exercise and coordinative exercise from the "Eastern exercise" perspective, (4) social interaction exercise, and (5) cool-down and meditation.
  Arms: Integrated Intervention Group (IIG)
Behavioral: Control Group — The Control Group is informed to maintain their lifestyles and invited to attend one 60-min online educational course per week. The participants are required to provide their physical activity behavior once every month for 6 months (6 times).
  Arms: Control Group

SUMMARY:
The current project is a single-blinded, double-arm, 6-month randomized controlled trial aiming to assess the effects of a integrated intervention program on neurocognitive function with respect to event-related potential in adults aged 45-70 years. Additionally, the potential impacts of apolipoprotein epsilon-4 alleles and the brain-derived neurotrophic factor will be explored.

DETAILED DESCRIPTION:
The current randomized clinical trial is designed to examine (1) whether a 6-month integrated intervention program (IIP) consisting of multiple exercise modalities, meditation, and social interaction could benefit neurocognitive function (e.g., inhibition) in middle-aged and older adults; (2) whether components of ERP will be influenced by the integrated intervention program; and (3) whether apolipoprotein E (ApoE) genotypes (ApoE e3/e4, ApoE e4/e4, ApoE e2/e2, ApoE e2/e3, ApoE e2/e4, and ApoE e3/e3), physical fitness, and brain-derived neurotrophic factor (BDNF) will influence the effects of an integrated intervention program on neurocognitive function and components of ERPs.

The study will randomly assign 100 eligible participants to either the IIP group or the control group in a 1:1 ratio. The IIP group will engage in 150 min of exercise per week, which consists of one 90-min on-site session and multiple online sessions, for 6 months. The control group will be invited to attend one 60-minutes online educational course per week for 6 months.

The neurocognitive function, the components of ERP, ApoE genotype, physical fitness, and BDNF will be assessed at the baseline (Baseline-Assessment) and the end of the 6-month intervention (Post-Assessment).

ELIGIBILITY:
Inclusion Criteria:

* Normal or corrected-to-normal vision
* Able to speak and read Chinese
* Scores of Mini-Mental Status Examination >= 25
* Physical Activity Readiness Questionnaire score < 0
* Able to conduct the exercise with moderate intensity
* Provide informed consent

Exclusion Criteria:

* Diagnosed or self-reported cognitive problems (e.g., mild cognitive impairment or dementia)
* Diagnosed or self-reported physical disease (e.g., untreated hypertension and chronic heart disease, stroke, brain tumor, musculoskeletal disorders, other exercise contradictions)
* Diagnosed or self-reported major psychiatric illness (e.g., major depression, schizophrenia)
* Diagnosed or self-reported neurodegenerative disease (e.g., Alzheimer's disease or other dementias, Parkinson's disease (PD) and PD-related disorders, Huntington's disease)
* History of alcohol or drug abuse
* History of chemotherapy
* Traveling consecutively for three weeks or more during the study
* Unwillingness to be randomized to one of the two groups
* Currently participating in another study trial

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Inhibition: Changes in Stroop test performance | 30 minutes each at the baseline and at month 6
  The computerized Stroop test is administrated to assess participants' inhibitory function, and the changes in Stroop test performance from baseline to end of the intervention (i.e., month 6) will be examined.
Changes in neuroelectrical activities | 60 minutes each at baseline and at month 6
  The neuroelectrical activities during the computerized cognitive tasks is recorded and analyzed using the Neuroscan system. Changes in the neuroelectrical activities from baseline to end of the intervention (i.e., month 6) will be examined.

SECONDARY OUTCOMES:
ApoE genotype | 5 minutes at baseline
  A 6 mL serum sample is drawn from the antecubital veins. Based on the genetic biomarkers (rs429358 and rs7412), participants' ApoE genotype is determined at the baseline.
Blood neurotrophic marker: Changes in brain-derived neurotrophic factor (BDNF) levels | 5 minutes each at baseline and at month 6
  A 6 mL serum sample is drawn from the antecubital veins to assess BDNF levels, and changes in BDNF levels from baseline to end of intervention (i.e., month 6) will be examined.
Physical fitness measurements: Changes in aerobic fitness | 30 minutes each at baseline and at month 6
  Participants' aerobic fitness is assessed using the submaximal cycle ergometer test, and changes in aerobic fitness from baseline to end of intervention (i.e., month 6) will be examined.
Physical fitness measurements: Changes in muscular fitness | 15 minutes each at baseline and at month 6
  Muscular fitness is assessed using either the push-up test/30 seconds or the chair stand test/30 seconds, and changes in muscular fitness from baseline to end of intervention (i.e., month 6) will be examined.
Physical fitness measurements: Changes in flexibility | 15 minutes each at baseline and at month 6
  Flexibility is assessed using the sit-and-reach test, and changes in flexibility from baseline to end of intervention (i.e., month 6) will be examined.
Psychosocial measures: Changes in mindfulness | 5 minutes each at baseline and at month 6
  Mindfulness level is assessed using the 15-items (1-6 Likert scale) Chinese version of the Mindful Attention Awareness Scale (MAAS) questionnaire. Higher mean scores of the 15 items indicate higher levels of dispositional mindfulness. Changes in mindfulness scores from baseline to end of intervention (i.e., month 6) will be examined.
Psychosocial measures: Changes in depression | 5 min each at the Baseline-Assessment and at the Post-Assessment
  Geriatric Depression Scale (GDS-15) is utilized to assess older adults' depression levels using 15 'Yes/No' items. Scores between 5 and 9 indicate mild symptoms, and a score of 10 and above indicates moderate symptoms. Changes in depression from baseline to end of intervention (i.e., month 6) will be examined.
Psychosocial measures: Changes in sleeping quality | 5 minutes each at baseline and at month 6
  The Chinese version of the Pittsburgh Sleep Quality Index will be used to assess individual's general sleep quality over a 1-month time interval. Participants complete 9 questions, and lower scores reflect better sleep quality. Changes in sleep quality from baseline to end of intervention (i.e., month 6) will be examined.
Psychosocial measures: Changes in health-related quality of life | 10 minutes each at baseline and at month 6
  Health-related quality of life via the 24-items (1-5 Likert scale) WHOQOL-OLD-Taiwan is used to measure the quality of life in older persons. The higher scores indicate better quality of life. Changes in health-related quality of life from baseline to end of intervention (i.e., month 6) will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Kai Chang, PhD, Principal Investigator — Department of Physical Education and Sport Sciences, National Taiwan Normal University
Locations (2):
- Taiwan (2):
  - Yu-Kai Chang, Taipei
  - Yu-Kai Normal Chang, Taipei

IPD SHARING:
Plan to Share IPD: No